CLINICAL TRIAL: NCT02243956
Title: Food Design for Improved Cognitive Performance/Effects on Cognitive Functions and Mood of Food Products Rich in Polyphenols
Brief Title: Effects on Cognitive Functions and Mood of Food Products Rich in Polyphenols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Anti-Diabetic Food Centre (Other)
Responsible Party: Principal Investigator, Anne Nilsson, PhD, Associate Professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AFC-2013/619
Record Dates: First submitted 2014-09-10; First posted 2014-09-18 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Cognitive Performance; Mood; Cardiometabolic Risk Markers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flavanol rich food product (Experimental): A portion of a common flavanol rich food product is consumed daily for 4 weeks
  Interventions: Other: Flavanol rich food product
- Non-flavanol food product (Placebo Comparator): A portion of a product similar to the experimental Product, but instead contains low amounts of flavanol, is consumed Daily for 4 weeks as a control.
  Interventions: Other: Flavanol rich food product

INTERVENTIONS:
Other: Flavanol rich food product — polyphenol rich test product

SUMMARY:
The purpose of this study is to investigate effects of a selected food product rich in polyphenol on cognitive performance and mood.

DETAILED DESCRIPTION:
The metabolic syndrome (MetS) includes a cluster of dysfunctions that identifies subjects at risk of developing type-2 diabetes and cardiovascular disease (CVD). A key feature appears to be chronic increased inflammation and activation of the innate system. Consequently, increased low-grade inflammation has been connected to adverse effects on insulin sensitivity, glucose- and lipid metabolism, and blood pressure, and circulating markers of inflammation such as IL-6. A growing body of evidence also link low-grade inflammation to poorer cognitive functioning. Type 2 diabetes, MetS, and glucose intolerance are increasingly being associated with impaired cognition.

Dietary patterns which promote sub-clinical inflammation are increasingly being considered predictive of future risk of CVD and type-2 diabetes. Epidemiological data shows that a high consumption of vegetables and fruits is associated with a lowered risk of cancer and cardiovascular disease, which may be due to the high concentrations of polyphenols or other anti-oxidants that are found in such foods.

In the presently described project it is hypothesized that four weeks daily consumption of a product specific high in flavanols can improve metabolic risk variables and cognitive functions in healthy subjects.

The purpose is therefore to investigate effects of flavanols on cognitive functions and cardiometabolic risk, and to investigate relations between cardiometabolic risk markers and cognitive performance. The test product is a commonly used food product, known to be specifically rich in flavanols. The effects of the test product is compared with effects of a control product that is based on a similar food product but is lacking flavanols.

Test parameters:

Cognitive tests: Working memory tests (an oral test), selection attention test (measure also reaction time, a computerized test ), and stroop test (a computerized test.

Mood is determined for 6 different mood sensations using VAS scales.

Bio markers in blood: glucose regulation (glucose, insulin), markers of inflammation and oxidative stress (IL-6, MDA, oxLDL), blood lipids (total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides), vascular function (P-Selectin, PAI-1, NO), gut hormones involved in metabolism and satiety (PYY, GLP-1) gut hormon involved in mucosa integrity (GLP-2), markers of brain function (BDNF, neurotensin).

Blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and men
* Between 50-70 years
* BMI 19-25

Exclusion Criteria:

* Metabolic diseases
* Food allergies
* Smoker

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
working memory (WM) capacity | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, working memory capacity is determined four times in the postprandial phase up to 3.5h after breakfast.
  The test food product or control is consumed fasting, and after 30 min a standardised breakfast is served. WM tests are performed at 60 min, 120 min, 165 min and 210 min after commencing the intake of test Product. One test takes approximately 8 min to carry out.

SECONDARY OUTCOMES:
mood assessment | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, subjects registered mood sensations at fasting and five times in the postprandial phase up to 3,5h after breakfast.
  Self-reported sensations of mood and feelings of activation was assessed with a modified bipolar variant of the Swedish Core Affect Scales (SCAS) comprising six rating scales of two orthogonal dimensions of core affect: valence (unpleasantness-pleasantness) and activation (quietness-excitement).
  Mood scales are filled out at fasting, prior to the standardised breakfast served after 30 min and directly after cognitive tests started at 60 min, 120 min, 165 min and 210 min after commencing the intake of test product.

OTHER OUTCOMES:
blood pressure | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, blood pressure is determined at fasting and four times in the postprandial phase up to 3,5h after breakfast.
  Blood pressure is determined at fasting and at 60 min, 90 min, 150 min and 180 min, prior to other test variables collected at the same test Point.
glucose regulation | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, blood glucose is determined fasting and then eight times in the postprandial phase up to 3.5h after the standardised breakfast
  Blood glucose concentrations (determined in capillary blood), and insulin (determined in venous blood). Blood tests are collected repeatedly during 3h after a standardised breakfast consumed 30 min after commencing the test product/Control Product.
selective attention (SA) | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, selective attention is determined three times in the postprandial phase up to 3.5h after the standardised breakfast
Vascular function | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, vascular marker is determined fasting and up to 3.5h after the standardised breakfast
Blood lipids | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, blood lipids are determined fasting and up to 3.5h after the standardised breakfast
Marker of inflammation | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, inflammatory markers in blood are determined fasting and up to 3.5h after the standardised breakfast
Markers of oxidative stress | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, markers of oxidative stress are determined in blood at fasting and then up to 3.5h after a standised breakfast
Gut peptides | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, gut peptides are determined in blood at fasting
markers of brain function | Each of the two intervention periods is 4 weeks. At the first and last day in each intervention periods, markers of brain finction are determined in blood at fasting
Stroop test | Each of the two intervention periods is 4 weeks. At the first and last day Stroop tests are performed three times after a standardised breakfast up to 3,5h .

CONTACTS AND LOCATIONS:
Locations (1):
- Lund Univercity, Medicon village, Functional Food Science Centre, Lund, Sweden